CLINICAL TRIAL: NCT05976607
Title: Linical Study of 18F Labeled Probe Targeting Fibroblast Activating Protein and Integrin avβ3 (FAPI-RGD) in Renal Tumors
Brief Title: Clinical Study of 18F -FAPI-RGD in Renal Tumor
Status: Completed | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Wang, Principal Investigator, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPH- renal tumor
Record Dates: First submitted 2023-07-26; First posted 2023-08-04 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Renal Tumor
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about the value of 18F-FAPI-RGD PET/CT imaging in Renal Tumor. Participants will undergo clinical evaluation and 18F-FAPI-RGD PET/CT examination.

DETAILED DESCRIPTION:
Early detection, accurate diagnosis and staging are the keys to effective treatment of kidney cancer patients.Pathological diagnosis is still the gold standard, but renal perforation is invasive examination, there are certain complications, the most common is bleeding and hematoma, rare renal arteriovenous fistula formation and infection.A non-invasive test with high accuracy is expected.68Ga-FAPI-04 has been reported to be superior to 18F-FDG in the study of bone metastases in RCC patients, and in addition to detecting more metastases than 18F-FDGPET/CT, uptake is 3-4 times higher than 18F-FDG.There are also many literatures reporting that APIPET/CT may be better than 18F-FDGPET/CT in the detection of various malignant tumors, and FAPI targeted imaging is a promising way in the diagnosis and treatment of papillary renal cell carcinoma.

18F-FPPRGD2PET/CT may be a useful tool for monitoring early response to anti-angiogenic therapy in patients with mRCC.18F-FPRGD2PET/CT reliably estimated the expression of integrin αvβ3 in renal tumors, and in clear cell RCC(ccRCC) groups, 18F-FPRGD2PET signal correlated with the expression of integrin αvβ3 in tumor cells.In the papillary RCC(pRCC) group, the signal was correlated with the expression of αvβ3.The expression of integrin αvβ3 in ccRCC cells was significantly higher than that in pRCC cells.These findings are consistent with results obtained with other RGD-based tracers in various cancers.The expression level of integrin αvβ3 in tumor cells is associated with invasiveness and metastasis potential, and quantifying it with PET may contribute to the study of integrin αvβ3 as a prognostic factor.

Heterodimer peptide FAPI-RGD was synthesized from FAPI and RGD.FAPI-RGD is a heterodimeric peptide that targets FAP and αvβ3-integrin receptors, 68Ga-FAPI-RGDPET/CT imaging has been used in clinical imaging studies of patients with various tumors.So, we plan to use 18F-FAPI-RGD PET/CT imaging is used in the diagnosis and treatment of renal cancer, and preliminary experiments have confirmed that this examination has a good imaging effect.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* No gender difference
* Patients who have been diagnosed with, or are clinically highly suspected of, renal tumors and have had no other treatment within 3 months

Exclusion Criteria:

* Patients with a second primary tumor
* Pregnant or breastfeeding
* Severe liver or kidney disease
* Claustrophobia or other PET/CT scan contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed or highly suspected Renal Tumor
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Correlation between clinical indicators and PET/CT results | 2 months
  Correlation of Clinical immunohistochemical indexes, ultrasound, enhanced CT, MRI, laboratory examination indexes and 18F-FAPI-RGD PET/CT results

CONTACTS AND LOCATIONS:
Locations (1):
- Departments of Nephrology, Sichuan Provincial People's Hospital, Chengdu, Sichuan, China